CLINICAL TRIAL: NCT01722565
Title: Randomized, Controlled, Prospective Study of the Use of a Mesh to Prevent Parastomal Hernia After Laparoscopic Abdominoperineal Resection
Brief Title: Prospective Study of the Use of a Mesh to Prevent Parastomal Hernia After Laparoscopic Abdominoperineal Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LAP-APR-2012-028
Record Dates: First submitted 2012-11-04; First posted 2012-11-07 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernias; Tolerance of lightweight meshes; laparoscopic abdominoperineal resection
MeSH Terms: interventions — Polypropylenes; glycolide E-caprolactone copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesh Group (Experimental): Patients receiving conventional sigmoid end colostomy plus a preperitoneal lightweight mesh Physiomesh® by laparoscopic procedure
  Interventions: Procedure: laparoscopic abdominoperineal resection with a lightweight mesh (polypropylene and poliglecaprone 25)
- Control Group (No Intervention): Patients receiving conventional sigmoid end colostomy by laparoscopic procedure, without mesh

INTERVENTIONS:
Procedure: laparoscopic abdominoperineal resection with a lightweight mesh (polypropylene and poliglecaprone 25)
  Arms: Mesh Group

SUMMARY:
Introduction: parastomal hernia (PH) is a frequent complication after an ostomy, despite the many prevention and treatment techniques that have been described. Since the introduction of laparoscopy, the frequency of PH is even higher than in open surgery. This type of hernia remains a surgical problem of considerable importance, requiring significant consumption of public health and economic resources, and representing a major alteration of the quality of life of these patients.

Objective: to evaluate the effectiveness of the insertion of a prosthesis to prevent PH in elective surgery for laparoscopic abdominoperineal resection.

Methodology: prospective, multidisciplinary, multi-center randomized controlled study. Control group: Rectal neoplasms undergoing elective surgery for laparoscopic abdominoperineal resection. Study group: Rectal neoplasms undergoing elective surgery for laparoscopic abdominoperineal resection with a lightweight mesh (polypropylene and poliglecaprone 25). Sample size was calculated based on a proportion of parastomal hernia of 65% in the control group and 15% in the study group. With an α risk =0.05 and 1- β= 0.8, 28 patients are required, 14 per group. Estimating a drop-out rate of 10%, the final number will be 32 patients. The efficacy will be evaluated clinically at six months and abdominal CT will be performed at 12 months along with another clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex intervened electively for colorectal surgery (rectal cancer) in whom definitive colostomy is indicated after laparoscopic abdominoperineal amputation.
* Life expectancy above 12 months

Exclusion Criteria:

* - Patients with allergy or intolerance of the compounds in the mesh
* Carriers of prosthetic meshes in the area of the ostomy
* Patients electively intervened for colorectal surgery (neo de reco) in whom definitive colostomy is indicated after abdominoperineal amputation but not via a laparoscopic approach.
* Cirrhotic patients
* Patients with life expectancy below 12 months due to underlying disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The reduction in the incidence of Parastomal Hernia after the mesh placement | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD, Principal Investigator — Corporacion Sanitaria Universitaria Parc Tauli; Manuel Lopez-Cano, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Corporacion Sanitaria Universitaria Parc Tauli, Sabadell, Barcelona, Spain